CLINICAL TRIAL: NCT05511389
Title: A Randomized Controlled Trial of Anterior-posterior Versus Anterior-lateral Shock Vectors for Electrical Cardioversion of Atrial Fibrillation
Brief Title: Anteroposterior Versus Anterolateral Electrode Position for Electrical Cardioversion of Atrial Fibrillation
Acronym: SHOCK-VECTOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Omar Ibrahim, Adult Cardiology Fellow, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14093
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Intervention Model Description: With a partial factorial randomization to manual pressure versus not (second intervention) if the first randomized attempt is unsuccessful at restoring normal heart rhythm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterolateral shock vector (Active Comparator): Patients with electrodes placed on the chest to obtain an anterolateral (front-to-side placement; also known as anteroapical) shock vector.
  If first shock is unsuccessful, participants who proceed to a second shock will be randomized to manual pressure versus none but electrode placement will remain the same.
  Interventions: Other: Anterolateral electrode position; Other: Manual pressure
- Anteroposterior shock vector (Active Comparator): Patients with electrodes placed on the chest to obtain an anteroposterior (front-to-back placement) shock vector.
  If first shock is unsuccessful, participants who proceed to a second shock will be randomized to manual pressure versus none but electrode placement will remain the same.
  Interventions: Other: Anteroposterior electrode position; Other: Manual pressure

INTERVENTIONS:
Other: Anterolateral electrode position — As described previously
  Arms: Anterolateral shock vector
Other: Anteroposterior electrode position — As described previously
  Arms: Anteroposterior shock vector
Other: Manual pressure — Manual pressure applied to the anterior electrode

SUMMARY:
Atrial fibrillation is the most common heart rhythm disorder (arrhythmia) worldwide. Nearly 40 million people are affected by atrial fibrillation worldwide, and this number is expected to increase by over 50% by 2050. Atrial fibrillation can cause strokes, heart attacks, heart failure, poor quality of life and even death. Almost half a million deaths worldwide are expected to be related to atrial fibrillation by 2050, and many billions of dollars are spent on atrial fibrillation related healthcare in North America every year.

We believe health outcomes for patients with atrial fibrillation, and healthcare costs associated with treating atrial fibrillation could be improved by optimizing existing treatments for atrial fibrillation and maximizing the likelihood of restoring normal heart rhythm. This allows them to benefit from lower stroke risk, better heart function, fewer symptoms and increased quality of life. Restoring normal sinus rhythm earlier prevents atrial fibrillation from causing permanent structural damage to the heart that in turn, makes atrial fibrillation intractable. Furthermore, patients in whom initial attempts to control atrial fibrillation are unsuccessful frequently require more medications or invasive catheter ablation procedures which are costly and carry substantial risk.

Electrical cardioversion is the main way physicians restore normal heart rhythm. In this procedure, the heart is "shocked" back into normal rhythm using two electrodes on the chest. Done correctly, this procedure is safe and effective. Many things are known about electrical cardioversion, for example, the best type and amount of electricity to use. What we don't know is the best position of the electrodes on the chest and whether applying direct, physical pressure to the electrodes makes cardioversion more successful. Our prior research suggests that improving positioning and applying pressure may improve cardioversion, but this finding needs to be verified with a rigorous, dedicated trial.

This study will demonstrate whether front-to-back, or front-to-side placement of the electrodes is more effective for electrical cardioversion of atrial fibrillation. We will also demonstrate whether manually applying pressure to the electrodes makes cardioversion more effective. Should our trial demonstrate a benefit for these techniques, we expect them to be universally applied around the world. Because hundreds of thousands of cardioversions are done each year, even small increases in cardioversion success means thousands fewer patients progress to needing more medications or invasive procedures to manage their atrial fibrillation.

We will study consenting adults presenting for non-urgent cardioversion of their atrial fibrillation. After explaining the study to participants and gaining their consent, we will randomly assign them to front-to-side or front-to-back electrode placement. Patients who remain in atrial fibrillation after the first shock will randomly receive either manual pressure or not. We will compare the success of cardioversion for front-side versus front-back electrode placement, and for manual pressure versus none. We will evaluate success by using electrocardiograms to assess for restoration of the heart rhythm back to normal.

We hypothesize that anterolateral electrode positioning is superior to anteroposterior electrode positioning. We also hypothesize that manual pressure is effective relative to none, when applied in patients who have had one unsuccessful shock already.

ELIGIBILITY:
Inclusion Criteria:

Consenting adult patients scheduled for non-emergent electrical cardioversion of Atrial Fibrillation or Flutter

Exclusion Criteria:

1. Insufficiently anticoagulation for cardioversion as per Canadian Cardiovascular Society guidelines or have not undergone trans-esophageal echocardiography to rule out left atrial thrombus
2. Anatomic contraindication to anterolateral or anteroposterior placement (e.g. skin conditions or wounds)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
First-shock cardioversion success | At time of intervention
  Reversion to sinus rhythm (5 consecutive P waves within 5 seconds of shock)

SECONDARY OUTCOMES:
Cumulative cardioversion success for anterolateral versus anteroposterior placement afte | At time of intervention
  Reversion to sinus rhythm (5 consecutive P waves within 5 seconds of shock)
Second shock success for manual pressure versus none | At time of intervention
  Reversion to sinus rhythm (5 consecutive P waves within 5 seconds of shock)

OTHER OUTCOMES:
Descriptive analysis of techniques and results for third, unrandomized, clinician directed shock | At time of intervention
  Reversion to sinus rhythm (5 consecutive P waves within 5 seconds of shock)
First shock cardioversion success (subgroup analysis) by electrode position | At time of intervention
  As above; exploratory subgroup analysis of: Males vs females, BMI > 30 vs BMI < 30, First episode atrial fibrillation versus recurrent, Duration of current episode >30 days vs <30 days, Left ventricular ejection fraction > 40% vs <40%, Left atrial volume index >34ml/m2 vs not, Premedication with amiodarone , sotalol or class 1 antiarrhythmic drugs versus not, History of cardiac surgery versus not
Second shock cardioversion success by manual pressure versus none | At time of intervention
  As above; exploratory subgroup analysis of: Males vs females, BMI > 30 vs BMI < 30, First episode atrial fibrillation versus recurrent, Duration of current episode >30 days vs <30 days, Left ventricular ejection fraction > 40% vs <40%, Left atrial volume index >34ml/m2 vs not, Premedication with amiodarone , sotalol or class 1 antiarrhythmic drugs versus not, History of cardiac surgery versus not
Total number of shocks by electrode positioning | At time of intervention
  Reversion to sinus rhythm (5 consecutive P waves within 5 seconds of shock)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Hamilton Health Sciences, Hamilton, Ontario
  - St Joseph's Healthcare Hamilton, Hamilton, Ontario